CLINICAL TRIAL: NCT03834142
Title: Pilot Study to Investigate the Feasibility and Tolerability of the Use of NSS-2-BRIDGE Device for Post-Operative Pain in Total Knee and Hip Arthroplasties, Bariatric, and Kidney Transplant Surgeries
Brief Title: NSS-2-BRIDGE Study for Total Knee and Hip Arthroplasties, Bariatric, and Kidney Transplant Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19020023
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Acute Pain; Arthropathy of Knee; Arthropathy of Hip; Pain, Postoperative; Kidney Transplant Donor; Bariatric Surgery Candidate
Keywords: Auriculotherapy; Pain Therapy
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: 10 subjects will be recruited in each surgical population (hip/knee, kidney, bariatric) to equal 30 total active participants. This will be compared to 10 controls in each surgical population, for a total of 60 participants in the entire pilot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): NSS-2-Bridge auricular therapy will be given in addition to standard of care.
  Interventions: Device: NSS-2 Bridge
- Control (No Intervention): No intervention, subject receives standard of care

INTERVENTIONS:
Device: NSS-2 Bridge — The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal.
  Arms: Intervention

SUMMARY:
The current opioid epidemic has led to a renewed interest in exploring non-pharmacological techniques to treat post-operative pain. An increasing number of patients are suffering from the adverse effects of opioid use following surgery, including post-operative nausea and vomiting, respiratory depression, immunosuppression, constipation, and most recently, addiction. In the United States, over $600 billion is spent every year on opioid addiction, including $79 billion related to opioid addiction following surgery. Despite many initiatives to decrease the use of opiates in the preoperative setting, opioids continue to be regularly prescribed before, during and after surgery. Although the risk of opioid addiction following surgery is recognized, the percentage of patients becoming addicted to opioids following surgery is not well understood. To date, there has been virtually no agreement regarding the duration and dosage that qualify for opioid dependence following surgery, nor that a clear estimation of the factors such as biological, psychosocial and socioeconomic that increase the risk of using opioids for extended periods of time after surgery. Therefore, in order to combat this growing health crisis at the ground level, it is incumbent upon the medical community to explore alternative methods of pain control to treat the surgical population in order to change the incidence of post-operative opioid addiction.

Percutaneous Nerve Field Stimulation (PNFS) is one of these recognized methods that ongoing research has shown to be effective as a complementary method of pain management. While PNFS is not a novel concept, clinical indications of auricular field stimulation have been limited in the past due to requirement of bulky, stationary and non-disposable stimulators and electrodes. These technological limitations made it difficult to establish the real clinical potential of auricular stimulation for the perioperative management of pain in surgical patients, despite the demonstration that auriculotherapy has been shown to relieve pain in the postoperative setting.

The NSS-2- BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal. These symptoms include pain, anxiety and post-operative nausea and vomiting; conditions which are also present following major orthopedic surgery such as knee and hip arthroplasties. The use of the NSS-2 BRIDGE device has been demonstrated to provide significant analgesia in patients with abdominal pain syndrome, and clinical trials are ongoing to assess the benefit of this approach for post-operative pain management. As compared to the present use of opioids for perioperative pain management, the use of a complementary, non-pharmacologic approach offers the advantage of analgesia without the associated side effects.

DETAILED DESCRIPTION:
An open-label, pilot study will investigate forty individuals, ten of which will be scheduled for total hip arthroplasty, ten will be scheduled for total knee arthroplasty, ten scheduled for kidney transplant and ten for bariatric surgery, will be approached and consented for this trial. Their data in regards to their post-operative pain, nausea, and analgesia use will be compared to 10 historic subjects who had the same surgeries in January (TKA/THA) or September (kidney transplant/bariatric) of 2019. The subjects who receive the NSS-2-BRIDGE will also be monitored for comfort with the device for the tolerability and feasibility of utilizing this device in the future to treat post-operative pain.

Once a patient has given and signed informed consent to participate in the study, demographic information and medical history will be collected from each participant on the day of the joint replacement/kidney transplant/bariatric surgery. Data will be de-identified and kept in a locked cabinet in a locked office. The PI and the research coordinator have been trained in placing the NSS-2-BRIDGE and will apply the device in the immediate post-operative setting (post-anesthesia care unit, PACU). The device will be attached behind the ear with double-sided tape. It contains three electrodes which will be applied to the ear and a ground which will be placed on the patient's lobe. Each electrode and the ground will be secured with adhesive bandages. The patient will be informed at the time of consent and after the implantation of the device that they can have the device removed any time after its application. Once the device is placed patients will be asked to perform a "pinch test" throughout the duration of their time wearing the device. To perform the "pinch test" they must pinch down on the electrodes and ground to ensure they are still placed in their designated locations and have not come loose.

As per standard of care, at 24, 48, 72, 96 and 120 hours post-operatively pain scores will be collected at rest and movement, total opioid consumption, as well as the devise tolerability. Additionally as per other pain pilot IRB approved projects, we shall also collect common medical information including time to bowel movement, PONV, time to oral intake (liquid and regular diet), time to hospital discharge, intensive care unit (ICU) admission, readmission to the hospital, readmission due to pain related issues, quality of recovery after joint replacement, overall patient satisfaction, and patient satisfaction related to pain management.

When the patient is discharged from the hospital, they will be asked to complete a patient satisfaction survey. If the patient should be discharged prior to 120 hours post-operatively, they will be asked to wear the device home. They will also be ask to remove the device at 120 hours (five days) after device placement and dispose of it in their home. We will provide removal instructions. Data post- hospital discharge regarding pain scores, opioid consumption, and device tolerability will be collected after discharge by calling the patient every day for 120 hr. following the placement of the device.

At UPMC Shadyside, we expect the patients undergoing primary unilateral either total hip or total knee surgery to be discharged on the day of surgery, or the next day but no later than 48 hrs following surgery. Therefore, for the patients in whom a Bridge device will be placed following surgery, it will be possible to document, if during the 120 hrs following the placement of the device, the patient returned to the hospital because of pain. This will be documented in the patient chart and therefore will be available for review.

Given that most post-bariatric patients are discharged at 72 hours or before, pain scores, opioid needs, and device tolerability at 96 and 120 hours will be collected from the patient by calling them after discharge. Participants will be called once daily up until day 5 and asked to report information. Phone calls to patients after discharge are consistent with routine clinical care. If the kidney transplant patient is discharged prior to 120 hours (5 days), they will also be called daily to record pain scores, opioid needs, and device tolerability for the time they are discharged up to 5 days post-device placement.

As stated in the protocol, each patient will be discharged according to the standard protocol defined by the surgical team. Data collected for both historical and study subjects will be the base of the standard clinical data collected for any patient undergoing surgery at UPMC SDY, UPMC Montefiore and UPMC MWH. After the patient is discharged from the hospital data related to pain, nausea and vomiting and opioid consumption will be obtained by a daily phone call.

The historical controls will include a medical chart review of patients from the Acute Perioperative Pain Service at UPMC Shadyside Hospital. Data collection includes total narcotic/non-opioid analgesic requirement, pain scores and nausea and vomiting after the surgery. Other information collected from the medical record will include age, race and medical history. Additionally, we will also collect common medical information including time to bowel movement, time to oral intake (liquid and regular diet), time to hospital discharge, intensive care unit (ICU) admission, readmission to the hospital, readmission due to pain related issues. No Personal Health Identifiers will be collected from the historical controls.

The subjects in whom the Bridge device will be placed will receive the same standard ERAS protocol as the patients who will be used as historical control.

No power analysis will be performed. However, the tolerability of the placement of the bridge device (focus of this study) will be assessed using the pain scores.

We will record pain scores before and after the placement of the Device (prior to leaving the recovering room, and at 24, 48, 72, 96 and 120 or until discharge from the hospital) and compare it to the historical data of pain scores recorded prior to discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Elective Total Knee OR Total Hip Arthroplasties OR Kidney transplant surgery OR Bariatric surgery

Exclusion Criteria:

* History of active depression, anxiety or catastrophizing
* Active alcoholism or drug abuse
* Severe chronic pain condition that requires daily preoperative opioid dependence
* History of hemophilia
* Patients with cardiac pacemakers or other implanted devices (e.g. vagal nerve simulators)
* Patients with psoriasis vulgaris diagnosis
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (3):
- United States (3):
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention-Kidney: NSS-2-Bridge auricular therapy will be given in addition to standard of care.
  NSS-2 Bridge: The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal.
- Control-Kidney: Subject receives standard of care
Period: Overall Study
Arm/Group | Intervention-Kidney | Control-Kidney
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Kidney Transplant Donor
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.7) | 42 (11.7) | 42.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of NSS-2 Bridge Device in Changing Perioperative Opioid Consumption
Description: Investigate the efficacy of the NSS-2 BRIDGE device in changing perioperative opioid consumption in opioid-naïve patients undergoing either a total hip or total knee arthroplasty procedure, bariatric or kidney donor surgeries. Since we are comparing to historical controls, we can only analyze data from when the controls were in the hospital. This could be within a 24hrs, 48hrs, 72 hours, 96 hours, or 120 hours timeframe.
Time Frame: This could be within a 24hrs, 48hrs, 72 hours, 96 hours, or 120 hours timeframe.
Population: Kidney Transplant Donor
Measure: Mean (Standard Deviation); unit: mg morphine equivalent (MME)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
mg morphine equivalent (MME) | 8.3 (9.6) | 33.5 (37.3)

2. Secondary Outcome: Pain Scores
Description: Investigate the efficacy of the NSS-2 BRIDGE device in changing perioperative NRS Pain scores in opioid-naïve patients undergoing either a total hip or total knee arthroplasty, bariatric or kidney donor surgeries. Since we are comparing to historical controls, we can only analyze data from when the controls were in the hospital.
  Numerical Rating Scale (NRS) Pain scores on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. higher scores represent a worse outcome.
Time Frame: Day of Surgery, 24 hours post-operative, 48 hours post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention-Kidney | Control-Kidney
Number analyzed (Participants) | 10 | 10
units on a scale
  Post-op 24 hour Pain Scores | 2.5 (2.0) | 6 (1.4)
  Post-op 48 hour Pain Scores | 1.6 (1.6) | 6.0 (2.8)

3. Secondary Outcome: Number of Participants With Post-operative Complications
Description: Investigate the number of participants that experienced post-operative complications .
Time Frame: Day of Surgery through post-operative day 5
Measure: Number; unit: Participants
Arm/Group | Intervention-Kidney | Control-Kidney
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

4. Secondary Outcome: Level of Comfort Wearing NSS-2 Bridge Device
Description: This was determined by asking the subject "How satisfied were you with the NSS-Bridge Device during the time in which it was worn, with 0 being the worst and 10 being the most satisfied?"
Time Frame: Post-operative day 5
Population: We were not able to reach 1 patient for the day 5 follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention - Kidney: NSS-2-Bridge auricular therapy will be given in addition to standard of care.
  NSS-2 Bridge: The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal.
Arm/Group | Intervention - Kidney
Number analyzed (Participants) | 9
units on a scale | 9 (3)

5. Secondary Outcome: Time to Hospital Discharge
Description: Length of time from end of surgery to discharge from hospital
Time Frame: Day of Surgery to post-op day 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention-Kidney | Control-Kidney
Number analyzed (Participants) | 10 | 10
days | 2.1 (2.9) | 2.2 (0.33)

6. Secondary Outcome: Time to Discharge From Recovery Room
Description: Length of time from end of surgery to discharge from the recovery room
Time Frame: Day of Surgery through post-operative day 5
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention-Kidney | Control-Kidney
Number analyzed (Participants) | 10 | 10
minutes | 134.9 (37.7) | 197.3 (152.5)

7. Secondary Outcome: Time to Oral Intake
Description: Length of time from end of surgery to first oral intake
Time Frame: Day of surgery to post-op day 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Intervention-Kidney | Control-Kidney
Number analyzed (Participants) | 10 | 10
hours | 5.3 (2.6) | 4.2 (2.7)

8. Secondary Outcome: Time to Ambulation
Description: Length of time from end of surgery to first ambulation
Time Frame: Day of surgery to post-op day 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Intervention-Kidney | Control-Kidney
Number analyzed (Participants) | 10 | 10
hours | 11.6 (7.4) | 18.9 (6.9)

ADVERSE EVENTS:
Time Frame: Day of surgery through 5 days post-op
Groups:
- Control-Kidney: No intervention, subject receives standard of care
Arm/Group | Intervention-Kidney | Control-Kidney
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03834142/Prot_001.pdf